CLINICAL TRIAL: NCT07072936
Title: Evaluation Of The Effect Of Mediterranean Diet On Serum Zonulin Levels And Treatment Success In Women Infertility
Brief Title: Effect Of The Mediterranean Diet On Zonulin And Infertility
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: SINEM BAYRAM (Other)
Responsible Party: Sponsor-Investigator, SINEM BAYRAM, Assoc. Prof., Baskent University
Organization: Baskent University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SINEM BAYRAM
Record Dates: First submitted 2025-01-20; First posted 2025-07-18 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-01

CONDITIONS: Infertility Female; Zonulin; Intestinal Permeability; Mediterranean Diet
Keywords: female infertility; serum zonulin; mediterranean diet; clinical pregnancy
MeSH Terms: conditions — Infertility, Female | interventions — Diet, Mediterranean

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- mediterranean diet group (Experimental): this group will apply mediterranean diet for 8 weeks
  Interventions: Behavioral: mediterranean diet
- control group (No Intervention): this group will apply routine diet for 8 weeks

INTERVENTIONS:
Behavioral: mediterranean diet — All questions of the intervention group, in which behavioural change was expected, were answered by the dietitian throughout the study and compliance with the diet was monitored with food consumption records.
  Arms: mediterranean diet group

SUMMARY:
The goal of this clinical trial is to learn if mediterranean diet works to treat infertility in women. It will also learn about the initial and end of study zonulin levels of mediterranean diet and control group. The main questions it aims to answer are:

* Does mediterranean diet lower the serum zonulin levels of participants?
* Does mediterranean diet improves the treatment success of participants with infertility? Researchers will compare mediterranean to a control group to see if diet works to treat infertility.

Participants will:

* Apply Mediterranean diet or routine diet without energy restriction for 8 weeks
* Visit the clinic once every 4 weeks for checkups and tests

ELIGIBILITY:
Inclusion Criteria:

* Being in the range of 18.5-29.9 kg/m2 BMI
* Having started infertility treatment

Exclusion Criteria:

* Having a chronic disease (diabetes mellitus, hypertension, etc.)
* Previous ovarian surgery
* Being diagnosed with PCOS, endometriosis
* Known autoimmune disease
* Thyroid disease

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Women (research focussed on female infertility)
Enrollment: 22 (Actual)
Dates: Start 2024-02-10 (Actual); Primary Completion 2024-05-20 (Actual); Study Completion 2024-08-30 (Actual)

PRIMARY OUTCOMES:
intestinal permeability | From enrollment to the end of treatment at 8 weeks
  serum zonulin levels

SECONDARY OUTCOMES:
infertility outcomes | From enrollment to the end of treatment at 8 weeks
  number of eggs collected
infertility outcomes | From enrollment to the end of treatment at 8 weeks
  number of embryos formed

CONTACTS AND LOCATIONS:
Locations (1):
- NovaArt, Ankara, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Data obtained through this study may be provided to qualified researchers with academic interest on infertility. Data or samples shared will be coded, with no PHI included. Approval of the request and execution of all applicable agreements (i.e. a material transfer agreement) are prerequisites to the sharing of data with the requesting party.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: Data requests can be submitted starting 9 months after article publication and the data will be made accessible for up to 24 months. Extensions will be considered on a case-by-case basis
Access Criteria: Access to trial IPD can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA)